CLINICAL TRIAL: NCT00866346
Title: A Phase I Study of PR1-Specific Cytotoxic T-Lymphocyte Infusion for Patients With Recurrent CML After Allogeneic Hematopoietic Transplantation
Brief Title: PR1-Specific Cytotoxic T-Lymphocyte Infusion With Recurrent Chronic Myelogenous Leukemia (CML) After Allogeneic Hematopoietic Transplantation
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study failed to accrue any patients due to regulatory issues with PR1 vaccine and T cell production.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0564; NCI-2012-01651 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-03-18; First posted 2009-03-20 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Chronic Myelogenous Leukemia
Keywords: Chronic Myelogenous Leukemia; CML; Allogeneic Hematopoietic Transplantation; Bone Marrow Transplant; PR1-Specific Cytotoxic T-Lymphocyte Infusion
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PR1-CTL (Experimental): Two infusions of PR1-specific T lymphocytes (donor immune cells) 60 days apart.
  Starting infusion dose 1 x 106 nucleated cells/kg.
  Interventions: Biological: PR1-primed lymphocyte (PR1-CTL) Infusion

INTERVENTIONS:
Biological: PR1-primed lymphocyte (PR1-CTL) Infusion — Two infusions of PR1-specific T lymphocytes (donor immune cells) 60 days apart.
  Starting infusion dose 1 x 106 nucleated cells/kg.
  Other Names: AHT; Allogenic Hemotopoietic Transplantation; PR1-CTL

SUMMARY:
Primary Objective:

To determine the maximally tolerated dose of donor PR1-specific cytotoxic T-lymphocytes (PR1-CTL) as treatment for relapsed or persistent chronic myelogenous leukemia (CML) after allogeneic hematopoietic transplantation from an HLA-matched related or unrelated donor.

Secondary Objectives:

1. To evaluate the immunological response following PR1-CTL treatment
2. To evaluate the clinical efficacy by determining clinical, cytogenetic and molecular response rates within 6 months

DETAILED DESCRIPTION:
Before treatment starts, you will have a complete physical exam, including blood (about 2 tablespoons) tests. You will have a chest x-ray and bone marrow will be collected. To collect a bone marrow sample, an area of the hip or chest bone is numbed with anesthetic and a small amount of bone marrow is withdrawn through a large needle. Women who are able to have children must have a negative blood pregnancy test.

You will be treated with donor immune cells (T lymphocytes) that will specifically target certain leukemia cells in your body. Each participant will receive two doses of donor cells, 60 days apart. The second dose will be given 60 days after the first dose, at a higher dose level, as long as no serious side effects occur after the first dose and there is still disease present. Four dose levels of PR1-specific T lymphocytes will be considered. Up to 30 patients will be treated in cohorts of 3, starting at the lowest dose level, and not skipping an untried dose level when escalating. The trial will be stopped early if the lowest dose level is found to be unacceptably toxic.

These cells will be given on an outpatient basis. After each donor cell infusions, you will be followed once a week in the outpatient clinic for at least 1 month and then every 3 months for at least one year. You will have routine blood (about 2 tablespoons) and urine tests at these visits. Participants experiencing side effects from their leukemia or leukemia treatment may need to be hospitalized earlier.

You will also receive several other medications to help decrease the risk of infections while your immune system is weak. These include preventative antibiotics, antiviral drugs, and antifungal drugs.

Bone marrow samples will be taken before the second cell infusion, and then 8 weeks, 12 weeks, 6 months and 1 year after the second cell infusion.

This is an investigational study. A total of up to 30 patients will be take part in this study. All will be enrolled at UTMDACC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic myelogenous leukemia (CML) who have previously undergone allogeneic hematopoietic transplantation and have evidence of disease, as defined by a,b or c (a) >5% Philadelphia chromosome positive cells on cytogenetic studies >/= 3 months post-transplant
2. (b) For patients in cytogenetic remission post-transplant, molecular evidence of disease at any time, defined as recurrence of quantitative PCR positivity for bcr-abl after achieving a molecular remission confirmed by 2 assays, 3 months apart or sooner if clinically indicated; OR a >10-fold increase in the relative expression of bcr-abl/abl detected and confirmed by a minimum of 2 consecutive PCR analysis, 3 months apart or sooner
3. (c) Molecular evidence of persistent disease on Real time PCR (bcr-abl/ abl x 100 of 0.05 and not declining) >3 months post-transplantation after treatment with imatinib mesylate.
4. Patients must have an HLA compatible related or unrelated donor capable of donating peripheral blood stem cells using apheresis techniques. This must be the same donor used for the original allogeneic hematopoetic transplantation. Patient must be HLA-A2 positive
5. ECOG performance status < or = 2
6. Serum bilirubin < or = 2 mg/dl
7. Serum transaminases < 4 x normal
8. Serum creatinine < or = 2 mg/dl
9. No active uncontrolled infection
10. HIV negative
11. No acute and/or chronic GVHD requiring systemic steroid therapy
12. Patient is not pregnant or breast feeding.
13. Signed informed consent
14. Patients must be off all immunosuppressive medications for at least 2 weeks prior to study entry.

Exclusion Criteria:

None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-03; Primary Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Maximally tolerated dose of donor PR1-specific cytotoxic T-lymphocytes (PR1-CTL) | Continuous reassessment, infusion day 0 and second infusion day 60+/- 7

CONTACTS AND LOCATIONS:
Overall Officials: Muzaffar H. Qazilbash, MD, Principal Investigator — UT MD Anderson Cancer Center; Richard E. Champlin, MD, BS, Study Chair — UT MD Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org